CLINICAL TRIAL: NCT06143696
Title: Study on the (Heart) Brain-gut Axis Mechanism of Qingxin Zishen Decoction in Treating Hot Flashes in Menopausal Syndrome Based on 16S rRNA Sequencing Technology
Brief Title: QXZS in Menopausal Syndrome Based on 16S rRNA Sequencing Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yun Chen (Other)
Responsible Party: Sponsor-Investigator, Yun Chen, Deputy Chief Physician, Jiangsu Province Hospital of Traditional Chinese Medicine
Organization: Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QXZS-Flora
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Menopause
Keywords: menopause; 16S rRNA; saliva flora; intestinal flora
MeSH Terms: interventions — femoston

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental group (Experimental): Qingxin Zishen decoction, oral administration, 1 dose a day, 2 times a day. For 28 days of medication, every 28 days. Observation time for 3 courses.
  Interventions: Drug: Qingxin Zishen decoction
- the control group (Active Comparator): Femoston, oral, 1 each time, once a day. For 28 days of medication, every 28 days. Observation time for 3 courses.
  Interventions: Drug: Femoston

INTERVENTIONS:
Drug: Qingxin Zishen decoction — Oral administration, 1 dose daily, twice a day
  Arms: the experimental group
Drug: Femoston — Oral administration, 1 pill each time, once a day
  Arms: the control group

SUMMARY:
The goal of this clinical trial is to explore the differences of intestinal flora and saliva flora between menopausal women, and the changes after medication, to find the association between the two and menopausal syndrome. The main questions it aims to answer are:

* What are the differences in intestinal flora and saliva flora in menopausal women with hot flashes and sweating.
* Whether these differences change after using traditional Chinese medicine and the association between intestinal, salivary flora and menopausal syndrome.

  60 patients will be screened according to the clinical experimental criteria. They will be randomly divided into trial group (30 cases) and control group (30 cases). The test group takes traditional Chinese medicine Qingxin Zishen decoction, and the control group takes oral Femoston, comparing the two groups with analysis of symptom improvement, intestinal flora and salivary flora with 16S rRNA sequencing technology.

ELIGIBILITY:
Inclusion Criteria:

* Those who meet the diagnostic criteria for menopausal syndrome and the TCM heart and kidney syndrome differentiation criteria.
* Women between the ages of 45~55.
* The score of the modified Kupperman Menopausal Symptom Rating Scale ≥ 15 points.
* Hot flashes and sweating≥ 3 times/day.
* Menopause ≥ 6 months.
* FSH > 10U/L during menopausal transition, 40U/L > after menopause, and estradiol (E2) < (10~20) pg/mL.

Informed consent, voluntary test. The process of obtaining informed consent should be in accordance with GCP regulations.

Exclusion Criteria:

* Other Chinese and Western drugs for the treatment of menopausal syndrome have been used after the onset of the disease.
* Have serious primary heart, liver, lung, kidney, blood or serious diseases that affect their survival.
* Contraindications to hormone therapy: known or suspected pregnancy; In perimenopausal women, menstrual disorders should be ruled out to exclude pregnancy-related problems such as intrauterine pregnancy, ectopic pregnancy, and trophoblastic disease. Unexplained vaginal bleeding: Causes of vaginal bleeding include neoplastic, inflammatory, iatrogenic, traumatic, and ovarian dysfunction, which should be carefully identified before perimenopausal menstrual disorders are treated with sex hormones. Known or suspected breast cancer. Known or suspected sex hormone-dependent malignancy. Active venous or arterial thromboembolic disease within the last 6 months. Severe hepatic and renal insufficiency.
* Those who are unable to give full informed consent due to intellectual or behavioral disabilities.
* Suspected or confirmed history of alcohol and drug abuse.
* Allergies, such as a history of allergies to two or more drugs or foods; or those who are known to be allergic to the ingredients of this medicine.
* Patients who are participating in clinical trials of other drugs.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
16s rRNA high-throughput sequencing of the gut flora | Baseline (Before treatment) and 12th weeks of treatment
  16s rRNA is a highly conserved gene segment in bacteria and archaea, together with some variability. Sequencing the 16S rRNA gene allowed us to identify different genera and species present in the microbial community and to assess their relative abundance.
16s rRNA high-throughput sequencing of the saliva flora | Baseline (Before treatment) and 12th weeks of treatment
  16s rRNA is a highly conserved gene segment in bacteria and archaea, together with some variability. Sequencing the 16S rRNA gene allowed us to identify different genera and species present in the microbial community and to assess their relative abundance.

SECONDARY OUTCOMES:
Hot flashes and sweating on a five-point scale. | Baseline (Before treatment) at the 4th, 8th and 12th weeks of treatment
  The symptoms of hot flashes and sweating were recorded as none, mild, moderate, severe, and very severe, and were recorded as 0, 1, 2, 3, and 4 points. The individual scores of the two groups before and after treatment at the end of the 4th, 8th and 12th weeks were compared.
Modified Kupperman rating scale | Baseline (Before treatment) at the 4th, 8th and 12th weeks of treatment
  The Kupperman Index (KMI) score was used to include 13 menopausal related symptoms such as vasomotor symptoms, paresthesias, insomnia, etc., and each symptom was divided into 0-3 points according to severity, and multiplied by different coefficients to obtain the menopausal symptom index, when the index > 35 indicates severe symptoms, 21-35 indicates moderate symptoms, and 15-20 indicates mild symptoms. The individual scores and total scores of the two groups before and after treatment at the 4th, 8th and 12th weekends were compared

CONTACTS AND LOCATIONS:
Locations (1):
- Yuxin Zhou, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No